CLINICAL TRIAL: NCT04661397
Title: A Single-Dose, Open-Label, Randomized, Replicate Crossover Pivotal Bioequivalence Study in Healthy Adult Participants to Assess the Bioequivalence of Darunavir 675 mg, Emtricitabine 200 mg, and Tenofovir Alafenamide 10 mg in the Presence of Cobicistat 150 mg When Administered as a Fixed Dose Combination (Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide) Compared to the Co-administration of the Separate Agents (Darunavir, Cobicistat, and Emtricitabine/Tenofovir Alafenamide), Under Fed Conditions
Brief Title: A Study in Healthy Participants to Assess the Effect of Darunavir, Emtricitabine, and Tenofovir Alafenamide in the Presence of Cobicistat as Fixed Dose Combination (Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide) Compared With Co-administration of the Separate Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108922; 2020-003396-18 (EudraCT Number); TMC114FD2HTX1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Darunavir; emtricitabine tenofovir alafenamide; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive Treatment A (a single dose of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide [D/C/F/TAF] as one fixed dose combination [FDC] tablet under fed condition on Day 1) as per assigned treatment sequence (Treatment sequence ABBA or BAAB). A wash out period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC; Drug: Darunavir; Drug: Emtricitabine/Tenofovir Alafenamide; Drug: Cobicistat
- Treatment B (Active Comparator): Participants will receive Treatment B (a single dose of Darunavir [DRV], Emtricitabine/Tenofovir Alafenamide [F/TAF] and Cobicistat [COBI] tablet under fed condition on Day 1) as per assigned treatment sequence (Treatment sequence ABBA or BAAB). A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC; Drug: Darunavir; Drug: Emtricitabine/Tenofovir Alafenamide; Drug: Cobicistat

INTERVENTIONS:
Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC — Participants will receive a single dose of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC tablet orally as per assigned treatment sequence.
  Other Names: TMC114/JNJ-48763364/JNJ-35807551/JNJ-63625328
Drug: Darunavir — Participants will receive a single dose of Darunavir orally as per assigned treatment sequence.
Drug: Emtricitabine/Tenofovir Alafenamide — Participants will receive a single dose of Emtricitabine/Tenofovir Alafenamide tablet orally as per assigned treatment sequence.
Drug: Cobicistat — Participant will receive a single dose of Cobicistat tablet orally as per assigned treatment sequence.

SUMMARY:
The purpose of the study is to evaluate the single-dose pharmacokinetics (PK) and pivotal bioequivalence of 3 compounds Darunavir (DRV), emtricitabine (FTC), and tenofovir alafenamide (TAF) in the presence of cobicistat (COBI) when administered as an fixed dose combination (FDC) (Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide [D/C/F/TAF]) compared to the co-administration as the separate commercial formulations (DRV and F/TAF and COBI), under fed conditions, in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index (BMI = weight/height^2) between 18.5 and 30.0 kilogram per meter square (kg/m^2) (extremes included), and body weight not less than 50 kilogram (kg)
* Must be healthy on the basis of physical examination, medical history, vital signs, and electrocardiogram (ECG) performed at screening (results must be available on Day -1). If there are abnormalities, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must be healthy on the basis of clinical laboratory test performed at screening (results must be available on Day -1). If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* A woman (of childbearing potential) must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test, 4 days or less before dosing of the first treatment period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after receiving the last dose of study drug

Exclusion Criteria:

* Has history or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease (including bronchospastic respiratory disease), diabetes mellitus, hepatic or renal insufficiency (for example, estimated creatinine clearance below less than [<] 90 milliliter per minute [mL/min] at screening), gastrointestinal disease (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Had one or more of the laboratory abnormalities at screening as outlined in the protocol by the Division of Acquired immunodeficiency syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events and in accordance with the normal ranges of the clinical laboratory
* Clinically significant abnormalities during physical examination, vital signs, or 12 lead ECG at screening or at admission to the study center as deemed appropriate by the investigator
* Has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 1 year before screening or positive test result(s) for alcohol and/or drugs of abuse (such as hallucinogens, barbiturates, opiates, opioids, cocaine, cannabinoids, amphetamines, methadone, benzodiazepines, methamphetamine, tetrahydrocannabinol, phencyclidine, and tricyclic antidepressants) either at screening or on Day 1 of each treatment period
* Has known allergies, hypersensitivity, or intolerance to Darunavir (DRV),Cobicistat (COBI), Emtricitabine (FTC), and/or Tenofovir Alafenamide (TAF), or any of their excipients
* Is a woman who is pregnant, or breast-feeding, or planning to become pregnant during this study or within 90 days after the last intake of study drug, or a woman of childbearing potential who is unwilling to use acceptable methods of contraception
* Has a history of hepatitis A antibody immunoglobulin M (IgM), hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for hepatitis A antibody IgM, HBsAg or anti-HCV at screening
* Has a history of human immunodeficiency virus type 1 or type 2 (HIV-1 or HIV-2) infection, or tests positive for HIV-1 or HIV-2 at screening
* Has had any contact with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive or coronavirus disease-19 (COVID-19) patients within the last 2 weeks prior to admission to the clinical research center

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Darunavir, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  Cmax is the maximum observed analyte concentration.
Area Under the Analyte Concentration-time Curve from time Zero to Last Quantifiable time (AUC[0-last]) of Darunavir, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  AUC(0-last) is the area under the analyte concentration-time curve from time zero to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.

SECONDARY OUTCOMES:
Area Under the Analyte Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Darunavir, Cobicistat, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the analyte concentration-time curve from time zero to last quantifiable time, C(last) is the last observed measurable concentration, and lambda(z) is elimination rate constant.
Cmax of Cobicistat | Up to 72 hours post-dose
  Cmax is the maximum observed analyte concentration of Cobicistat.
AUC(0-last) of Cobicistat | Up to 72 hours post-dose
  AUC(0-last) is the area under the analyte concentration-time curve from time zero to the time of the last measurable (non-BQL) concentration, calculated by linear-linear trapezoidal summation.
Number of Participants with Adverse Events (AEs) | Up to 9 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Van Hemelryck S, Van Landuyt E, Ariyawansa J, Vanveggel S, Palmer M. Bioequivalence of a Pediatric Fixed-Dose Combination Tablet Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Compared With Coadministration of the Separate Agents in Healthy Adults: An Open-Label, Randomized, Replicate Crossover Study. Clin Pharmacol Drug Dev. 2023 Nov;12(11):1060-1068. doi: 10.1002/cpdd.1293. Epub 2023 Jun 19. PMID 37335552